CLINICAL TRIAL: NCT04649216
Title: A Phase I, Single-Center, Open-Label Study Investigating the Excretion Balance, Pharmacokinetics (PK) and Metabolism of a Single Oral Dose of [14C]PCO371 and PK of an Intravenous (IV) Tracer of [14C]PCO371 in Healthy Male Subjects
Brief Title: Excretion Balance, PK and Metabolism of a Single Oral Dose of [14C]PCO371
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCO006EU
Record Dates: First submitted 2020-11-11; First posted 2020-12-02 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — PCO371

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mass Balance (Experimental): Subjects will receive a single oral dose of [14C]PCO371 Oral Solution.
  Interventions: Drug: [14C]PCO371
- Absolute Bioavailability and Mass Balance (Experimental): Subjects will receive a single oral dose of PCO371 capsules, followed by a single IV infusion of [14C]PCO371 over 10 min, starting 2 h post-oral dose.
  Interventions: Drug: PCO371; Drug: [14C]PCO371

INTERVENTIONS:
Drug: PCO371 — PCO371 Capsule
  Arms: Absolute Bioavailability and Mass Balance
Drug: [14C]PCO371 — [14C]PCO371 Oral solution
  Arms: Mass Balance
Drug: [14C]PCO371 — [14C]PCO371 Solution for infusion
  Arms: Absolute Bioavailability and Mass Balance

SUMMARY:
This is a Phase I single center, open-label, non-randomized study in healthy male subjects, designed to evaluate the mass balance recovery, PK, metabolism and absolute bioavailability of single oral doses of PCO371. It is planned to enroll 12 subjects, with 6 subjects in each of 2 study parts. Subjects in Part 1 will receive a single oral dose of [14C]PCO371 Oral Solution. Subjects in Part 2 will receive a single oral dose of PCO371 capsules, followed by a single intravenous infusion of [14C]PCO371 Solution for Infusion over 10 min, starting 2 h post-oral dose. The study parts may be dosed in any order for logistical reasons (e.g. Part 2 may be dosed before Part 1). No subject will be permitted to take part in both study parts.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Aged 40 to 60 years inclusive at the time of signing informed consent.
3. Body mass index (BMI) of 18.5 to 30.0 kg/m2 as measured at screening.
4. Must be willing and able to communicate and participate in the whole study.
5. Subjects must have regular bowel movements (i.e. average stool production of >=1 and <=3 stools per day).
6. Must provide written informed consent.
7. Must agree to adhere to the contraception requirements.
8. Subjects must regularly consume 2 or more units of alcohol per week.

Exclusion Criteria:

1. Subjects who have taken any experimental (non-approved) drug (including placebo) either within 90 days before the administration of the study drug, or 6 times the T1/2 of the experimental drug, whichever is longer.
2. Subjects who have previously been administered IMP in this study. Subjects are not permitted to be dosed in both Part 1 and Part 2 of the study.
3. Subjects who have been administered IMP in any 14C-labelled ADME in the last 12 months.
4. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years.
5. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study.
6. Subjects who do not have suitable veins for multiple venipunctures / cannulation as assessed by the investigator or delegate at screening.
7. Clinically significant abnormal clinical chemistry, hematology, coagulation or urinalysis as judged by the investigator at screening or admission.
8. Abnormal (outside of reference range) serum calcium or corrected calcium as measured at admission or screening.
9. Elevated (> 2.5 × upper limit of normal [ULN]) alkaline phosphatase at admission or screening. Subjects with Gilbert's syndrome or elevated (above the ULN) aspartate aminotransferase (AST), ALT or total bilirubin at admission or screening.
10. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results.
11. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of <60 mL/min using the Cockcroft-Gault equation.
12. Confirmed positive drugs of abuse test result.
13. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, immunologic, metabolism, endocrine, neurological or psychiatric disorder, as judged by the investigator, blood dyscrasia, risk factors for osteosarcoma as judged by the investigator.
14. Evidence or any history of active diseases that might affect calcium, bone metabolism, or calcium-phosphate homeostasis.
15. Use of anti-coagulants (e.g. heparins, warfarin, and thrombolytic agents), anti-platelet medications (e.g. argatroban and ticlopidine), nonsteroidal anti-inflammatory drugs and aspirin within 2 weeks (or within 6 times the T1/2 of the drug, whichever is longer) prior to study drug administration.
16. Subjects who have taken any inducers of CYP3A4, P glycoprotein (e.g. St. John's wort), or BCRP within 1 month prior to study drug administration, or taken any inhibitors of CYP3A4, P-glycoprotein, or BCRP (including herbal products, diets, and drinks e.g. tonic water) within 2 weeks prior to study drug administration (or within 6 times the T1/2 of the drugs mentioned above, whichever is longer).

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Mass balance data for [14C]PCO371 Oral solution in urine | 1 week
  Amount of total radioactivity excreted in urine(Ae(urine)) and Ae(urine) expressed as a percentage of the radioactive dose administered (%Ae(urine)), cumulative amount of total radioactivity excreted in urine (CumAe(urine)) and CumAe(urine)expressed as a percentage of the radioactive dose administered (Cum%Ae(urine)) following oral administration of [14C]PCO371 Oral Solution.
Mass balance data for [14C]PCO371 Oral solution in feces | 5 weeks
  Amount of total radioactivity excreted in feces(Ae(feces)) and Ae(feces) expressed as a percentage of the radioactive dose administered (%Ae(feces)), cumulative amount of total radioactivity excreted in feces (CumAe(feces)) and CumAe(feces)expressed as a percentage of the radioactive dose administered (Cum%Ae(feces)) following oral administration of [14C]PCO371 Oral Solution.
Mass balance data for [14C]PCO371 Oral solution in urine and feces combined | 5 weeks
  Amount of total radioactivity excreted in urine and feces combined(Ae(total)) and Ae(total) expressed as a percentage of the radioactive dose administered (%Ae(total)), cumulative amount of total radioactivity excreted in urine and feces combined (CumAe(total)) and CumAe(total)expressed as a percentage of the radioactive dose administered (Cum%Ae(total)) following oral administration of [14C]PCO371 Oral Solution.
Absolute bioavailability (F) for PCO371 | 1 week
  Time of maximum observed concentration for PCO371 and a metabolite in plasma and for total radioactivity in plasma and whole blood following oral administration of [14C]PCO371 Oral Solution

SECONDARY OUTCOMES:
Pharmacokinetic data for [14C]PCO371 Oral Solution; Tmax | 1 week
  Time of maximum observed concentration for PCO371 and a metabolite in plasma and for total radioactivity in plasma and whole blood following oral administration of [14C]PCO371 Oral Solution
Pharmacokinetic data for [14C]PCO371 Oral Solution; Cmax | 1 week
  Maximum observed concentration for PCO371 and a metabolite in plasma and for total radioactivity in plasma and whole blood following oral administration of [14C]PCO371 Oral Solution
Pharmacokinetic data for [14C]PCO371 Oral Solution; AUC(0-last) | 1 week
  Area under the curve from time 0 to the time of last measurable concentration for PCO371 and a metabolite in plasma and for total radioactivity in plasma and whole blood following oral administration of [14C]PCO371 Oral Solution
Pharmacokinetic data for [14C]PCO371 Oral Solution; AUC(0-inf) | 1 week
  Area under the curve from time 0 extrapolated to infinity for PCO371 and a metabolite in plasma and for total radioactivity in plasma and whole blood following oral administration of [14C]PCO371 Oral Solution
Pharmacokinetic data for [14C]PCO371 Oral Solution; T1/2 | 1 week
  Terminal elimination half-life for PCO371 and a metabolite in plasma and for total radioactivity in plasma and whole blood following oral administration of [14C]PCO371 Oral Solution
Pharmacokinetic data for [14C]PCO371 Oral Solution; Cmax ratio | 1 week
  Ratio of PCO371: total radioactivity and ratio of a metabolite: total radioactivity based on Cmax following oral administration of [14C]PCO371 Oral Solution
Pharmacokinetic data for [14C]PCO371 Oral Solution; AUC ratio | 1 week
  Ratio of whole blood: plasma total radioactivity based on Cmax following oral administration of [14C]PCO371 Oral Solution
Pharmacokinetic data for [14C]PCO371 Oral Solution; B:P Cmax ratio | 1 week
  Ratio of whole blood:plasma total radioactivity based on Cmax following oral administration of [14C]PCO371 Oral Solution
Pharmacokinetic data for [14C]PCO371 Oral Solution; B:P AUC ratio | 1 week
  Ratio of whole blood:plasma total radioactivity based on AUC following oral administration of [14C]PCO371 Oral Solution
Metabolite profiling of plasma, urine and feces | 1 week
  The chemical structure of each metabolite accounting for >=5% of circulating radioactivity in plasma and accounting for >=5% of the dose in the urine and feces
Intravenous pharmacokinetic data for [14C]PCO371 Solution for Infusion; C0 | 1 week
  Concentration at end of infusion of [14C]PCO371 and total radioactivity in plasma following oral dose of PCO371 capsules and intravenous infusion of [14C]PCO371 Solution for Infusion.
Intravenous pharmacokinetic data for [14C]PCO371 Solution for Infusion; AUC(0-last) | 1 week
  Area under the curve from time 0 to the time of last measurable concentration of [14C]PCO371 and total radioactivity in plasma following oral dose of PCO371 capsules and intravenous infusion of [14C]PCO371 Solution for Infusion.
Intravenous pharmacokinetic data for [14C]PCO371 Solution for Infusion; AUC(0-inf) | 1 week
  Area under the curve from time 0 extrapolated to infinity of [14C]PCO371 and total radioactivity in plasma following oral dose of PCO371 capsules and intravenous infusion of [14C]PCO371 Solution for Infusion.
Intravenous pharmacokinetic data for [14C]PCO371 Solution for Infusion; T1/2 | 1 week
  Terminal elimination half-life of [14C]PCO371 and total radioactivity in plasma following oral dose of PCO371 capsules and intravenous infusion of [14C]PCO371 Solution for Infusion.
Intravenous pharmacokinetic data for [14C]PCO371 Solution for Infusion; CL | 1 week
  Total body clearance calculated after a single IV administration of [14C]PCO371 in plasma following oral dose of PCO371 capsules and intravenous infusion of [14C]PCO371 Solution for Infusion.
Intravenous pharmacokinetic data for [14C]PCO371 Solution for Infusion; Vz | 1 week
  Volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single IV administration of [14C]PCO371 in plasma following oral dose of PCO371 capsules and intravenous infusion of [14C]PCO371 Solution for Infusion.
Oral pharmacokinetic data for PCO371 capsule; Tmax | 1 week
  Time of maximum observed concentration for plasma concentration of PCO371 and a metabolite following oral dose of PCO371 capsules and intravenous infusion of [14C]PCO371 Solution for Infusion.
Oral pharmacokinetic data for PCO371 capsule; Cmax | 1 week
  Maximum observed concentration for plasma concentration of PCO371 and a metabolite following oral dose of PCO371 capsules and intravenous infusion of [14C]PCO371 Solution for Infusion.
Oral pharmacokinetic data for PCO371 capsule; AUC(0-last) | 1 week
  Area under the curve from time 0 to the time of last measurable concentration for plasma concentration of PCO371 and a metabolite following oral dose of PCO371 capsules and intravenous infusion of [14C]PCO371 Solution for Infusion.
Oral pharmacokinetic data for PCO371 capsule; AUC(0-inf) | 1 week
  Area under the curve from time 0 extrapolated to infinity for plasma concentration of PCO371 and a metabolite following oral dose of PCO371 capsules and intravenous infusion of [14C]PCO371 Solution for Infusion.
Oral pharmacokinetic data for PCO371 capsule; T1/2 | 1 week
  Terminal elimination half-life for plasma concentration of PCO371 and a metabolite following oral dose of PCO371 capsules and intravenous infusion of [14C]PCO371 Solution for Infusion.
Mass balance data for [14C]PCO371 Solution for Infusion in urine | 1 week
  Cumulative amount of total radioactivity excreted in urine expressed as a percentage of the radioactive dose administered (Cum%Ae(urine)) and cumulative amount of [14C]PCO371 excreted in urine expressed as a percentage of the [14C]PCO371 dose administered (Cum%Ae([14C]PCO371 urine))
Mass balance data for [14C]PCO371 Solution for Infusion in feces | 5 weeks
  Cumulative amount of total radioactivity excreted in feces expressed as a percentage of the radioactive dose administered (Cum%Ae(feces)) and cumulative amount of [14C]PCO371 excreted in feces expressed as a percentage of the [14C]PCO371 dose administered (Cum%Ae([14C]PCO371 feces))
Safety data for PCO371; Adverse event monitoring | 6 weeks
  Incidence and severity of adverse events
Safety data for PCO371; Incidence of laboratory abnormalities | 6 weeks
  Incidence of laboratory abnormalities, based on clinical laboratory tests ( i.e. hematology, clinical chemistry, coagulation and urinalysis test results)
Safety data for PCO371; 12-lead ECGs (Ventricular Rate) | 6 weeks
  Abnormality in Electrocardiograms (ECGs) Interpretation based on Ventricular Rate
Safety data for PCO371; 12-lead ECGs (PR interval) | 6 weeks
  Abnormality in Electrocardiograms (ECGs) Interpretation based on PR interval
Safety data for PCO371; 12-lead ECGs (QRS Duration) | 6 weeks
  Abnormality in Electrocardiograms (ECGs) Interpretation based on QRS Duration
Safety data for PCO371; 12-lead ECGs (QT interval) | 6 weeks
  Abnormality in Electrocardiograms (ECGs) Interpretation based on QT interval
Safety data for PCO371; 12-lead ECGs (QRS Axis) | 6 weeks
  Abnormality in Electrocardiograms (ECGs) Interpretation based on QRS Axis
Safety data for PCO371; 12-lead ECGs (QTcF interval) | 6 weeks
  Abnormality in Electrocardiograms (ECGs) Interpretation based on QTcF interval
Safety data for PCO371; 12-lead ECGs (Rhythm) | 6 weeks
  Abnormality in Electrocardiograms (ECGs) Interpretation based on Rhythm
Safety data for PCO371; Vital signs (Systolic blood pressure) | 6 weeks
  Abnormality in Systolic blood pressure
Safety data for PCO371; Vital signs (Diastolic blood pressure) | 6 weeks
  Abnormality in Diastolic blood pressure
Safety data for PCO371; Vital signs (Heart Rate) | 6 weeks
  Abnormality in Heart Rate
Safety data for PCO371; Vital signs (Oral temperature) | 6 weeks
  Abnormality in Oral temperature
Safety data for PCO371; Presense of abnormalities in Physical examinations | 6 weeks
  Abnormality in Physical examination findings

CONTACTS AND LOCATIONS:
Overall Officials: Chugai Pharma Europe Ltd., Study Director — clinical-trials@chugai-pharm.co.jp
Locations (1):
- Quotient Sciences, Nottingham, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).